CLINICAL TRIAL: NCT03794661
Title: Evaluation of the Infinity Deep Brain Stimulation Electrode Screening Mode Tool
Acronym: EVIDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABT-CIP-10245
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Essential Tremor; Parkinson's Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Masking Description: Outcomes assessor will be masked to subjects' deep brain stimulation programming.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): Clinician programmer electrode screening mode tool
  Interventions: Device: Clinician programmer electrode screening mode tool

INTERVENTIONS:
Device: Clinician programmer electrode screening mode tool — Provides a standardized workflow to guide clinicians or trained healthcare providers through the deep brain stimulation monopolar review screening process
  Other Names: Informity tool

SUMMARY:
The objective of this clinical investigation is to characterize the clinical performance of Abbott's Clinician Programmer Electrode Screening Mode tool (InformityTM tool) in programming InfinityTM deep brain stimulation (DBS) systems for patients with Parkinson's disease (PD) or essential tremor (ET).

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm, multi-center, post-market clinical investigation designed to evaluate Abbott's Informity tool for Infinity DBS systems.

This clinical investigation will be conducted at up to 5 centers in the United States.

Up to 40 patients were intended to enroll in the study. However the study was stopped after enrolling 8 subjects at 3 sites.

Subjects participating in this clinical investigation will be followed for 6 months. The expected duration of enrollment is 6 months. The total duration of the clinical investigation is expected to be 18 months. The primary and secondary endpoints will be evaluated when all subjects have completed their 6 month follow-up visits

ELIGIBILITY:
INCLUSION CRITERIA

Parkinson's disease patients:

1. Patient must provide written informed consent prior to any clinical study related procedure.
2. Patient is 18 to 80 years of age.
3. Patient is diagnosed with Parkinson's disease for at least 4 years according to standard practice.
4. Patient is willing to maintain a constant dose of anti-Parkinson's disease medication indicated as best medical management for at least 1 month prior to study enrollment.
5. Patient is willing and able to comply with the follow-up schedule for the length of the study.
6. Patient has been implanted with an 8-channel directional Infinity deep brain stimulation system in the subthalamic nucleus (STN) within the last 12 months.
7. Patient has had stable deep brain stimulation programming settings for at least 1 month prior to study enrollment.

Essential tremor patients:

1. Patient must provide written informed consent prior to any clinical study related procedure.
2. Patient is 18 to 80 years of age.
3. Patient is diagnosed with essential tremor for at least 4 years according to standard practice.
4. Patient is willing to maintain a constant dose of anti-tremor medication indicated as best medical management for at least 1 month prior to study enrollment.
5. Patient is willing and able to comply with the follow-up schedule for the length of the study.
6. Patient has been implanted with an 8-channel directional Infinity deep brain stimulation system in the ventral intermediate (Vim) thalamus within the last 12 months.
7. Patient has had stable deep brain stimulation programming settings for at least 1 month prior to study enrollment.

EXCLUSION CRITERIA

1. Individuals unable to make the decision to participate in a clinical investigation on their own.
2. Patient is currently programmed with segmented electrodes, and cannot tolerate omnidirectional programming.
3. Patient is being evaluated for a lead revision.
4. Patient has untreated clinically significant depression.
5. Patient has dementia that interferes with their ability to co-operate or comply with study requirements or comprehend the informed consent, as determined by the investigator.
6. Patient abuses drugs or alcohol.
7. Patient is currently enrolled or plans to enroll in another concurrent study that may confound the results of this clinical investigation.
8. Patient has a confirmation of diagnosis of a terminal illness associated with survival <12 months.
9. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the patient's ability to participate in the clinical study or to comply with follow-up requirements, or impact the scientific soundness of the clinical study results.
10. Pregnant or nursing patients and those who plan pregnancy during the clinical study follow-up period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley White, Study Chair — Abbott; Binith Cheeran, Study Director — Abbott Medical Devices Neuromodulation
Locations (3):
- United States (3):
  - Albany Medical Center, Albany, New York
  - The University of Texas Health Science at San Antonio, San Antonio, Texas
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 8 subjects at 3 investigation sites. Of which seven subjects were diagnosed with Essential Tremor and one subject with Parkinson's Disease. The first subject enrollment was on June 26, 2019.
Period: Overall Study
Arm/Group | Single Arm
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Essential Tremor [Count of Participants; unit: Participants] | 7
Parkinson's Disease [Count of Participants; unit: Participants] | 1
Years of essential tremor symptoms [Mean (Standard Deviation); unit: years] — Population: Of the total 8 subjects enrolled, 7 subjects were diagnosed with Essential Tremor and 1 subject with Parkinson's Disease.
  years
    number analyzed (Participants) | 7
    (all) | 26 (16)
Years since initial diagnosis of essential tremor [Mean (Standard Deviation); unit: years] — Population: Of the total 8 subjects enrolled, 7 subjects were diagnosed with Essential Tremor and 1 subject with Parkinson's Disease.
  years
    number analyzed (Participants) | 7
    (all) | 16 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Therapeutic Window Size With Selected Contact at the Informity Programming Visit Compared to Baseline
Description: Therapeutic window was defined as the electrical current at which the side effect appeared minus the electrical current at which complete therapeutic benefit was obtained. The reported value is the range of current between first side effect appearance and complete therapeutic benefit. The 'Selected contact' is the therapeutic window for the contact configuration selected for the patient's programming. The 'best contact' is the therapeutic window for the contact configuration that showed the widest therapeutic window during Informity testing.
Time Frame: At Day 21 compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Arm/Group | Single Arm
Number analyzed (Participants) | 8
milliampere (mA)
  Baseline | 1.37 (1.48)
  Informity Programming | 1.80 (1.35)

2. Primary Outcome: Change in Therapeutic Window Size With Best Contact at the Informity Programming Visit Compared to Baseline
Description: as for outcome 1
Time Frame: At Day 21 compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Arm/Group | Single Arm
Number analyzed (Participants) | 8
milliampere (mA)
  Baseline | 1.37 (1.48)
  Informity Programming | 2.34 (1.29)

3. Primary Outcome: Change in Therapeutic Electrical Energy Delivered (TEED) With Selected Contact at the Informity Programming Visit Compared to Baseline
Description: TEED measures the total energy delivered by the deep brain stimulation system, and is represented as delivery over a set, arbitrary period of time. TEED is determined by the programmed stimulation parameters and measured system impedance. The 'Selected contact' is the contact configuration selected for the patient's programming. The 'best contact' is the contact configuration with the lowest TEED during Informity testing.
Time Frame: At Day 21 compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: microjoule (μJ)
Arm/Group | Single Arm
Number analyzed (Participants) | 8
microjoule (μJ)
  Baseline | 46.6 (30.2)
  Informity Programming | 65.6 (94.5)

4. Primary Outcome: Change in Therapeutic Electrical Energy Delivered (TEED) With Best Contact at the Informity Programming Visit Compared to Baseline
Description: as for outcome 3
Time Frame: At Day 21 compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: microjoule (μJ)
Arm/Group | Single Arm
Number analyzed (Participants) | 8
microjoule (μJ)
  Baseline | 46.6 (30.2)
  Informity Programming | 31.4 (23.9)

5. Secondary Outcome: Motor Symptom Evaluation for ET Subjects- Change in Fahn Tolosa Marin Tremor Rating Scale (FTM-TRS) Scores at 3 Months
Description: Change in Fahn-Tolosa-Marin tremor rating scale for ET subjects at 3-month follow-up visit compared to baseline. Fahn-Tolosa-Marin tremor rating scale scores are expressed as a percentage of the total score possible (range of 0% to 100%), and lower scores indicate less severe motor symptoms.
Time Frame: At 3 months compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 5
score on a scale
  Baseline | 20.6 (9.8)
  3 months | 19.6 (7.8)

6. Secondary Outcome: Motor Symptom Evaluation for ET Subjects- Change in Fahn Tolosa Marin Tremor Rating Scale (FTM-TRS) Scores at 6 Months
Description: Change in Fahn-Tolosa-Marin tremor rating scale for ET subjects at 6-month follow-up visit compared to baseline. Fahn-Tolosa-Marin tremor rating scale scores are expressed as a percentage of the total score possible (range of 0% to 100%), and lower scores indicate less severe motor symptoms.
Time Frame: At 6 months compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 5
score on a scale
  Baseline | 20.6 (9.8)
  6 months | 18.2 (10.2)

7. Secondary Outcome: Mean Quality of Life for Essential Tremor Subjects as Measured by the Quality of Life in Essential Tremor (QUEST) at Baseline
Description: Mean quality of life will be measured by the QUEST for ET subjects at baseline. The QUEST questionnaire consists of 30 items, which are rated from 0 to 4, corresponding to the frequency (from never to always). Those 30 items assess how tremor impacts a function or how it can be associated with feelings or attitudes. The 30 items contribute to five sub scales (number of items contributing to each scale in parentheses): Physical/ADL (9), Psychosocial (9), Communication (3), Hobbies/Leisure (3), and Work/Finances (6). The score on each sub scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. Maximal score of 100 indicates worse quality of life, while minimal score 0 corresponds to best quality of life.
Time Frame: At baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 7
score on a scale
  Communication | 7 (13)
  Work / Finance | 17 (23)
  Hobbies / Leisure | 35 (35)
  Physical | 36 (22)
  Psychosocial | 24 (14)

8. Secondary Outcome: Mean Quality of Life for Essential Tremor Subjects as Measured by the Quality of Life in Essential Tremor (QUEST) at 3 Months
Description: Mean quality of life will be measured by the QUEST for ET subjects at 3 months follow-up visit. The QUEST questionnaire consists of 30 items, which are rated from 0 to 4, corresponding to the frequency (from never to always). Those 30 items assess how tremor impacts a function or how it can be associated with feelings or attitudes. The 30 items contribute to five sub scales (number of items contributing to each scale in parentheses): Physical/ADL (9), Psychosocial (9), Communication (3), Hobbies/Leisure (3), and Work/Finances (6). The score on each sub scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. Maximal score of 100 indicates worse quality of life, while minimal score 0 corresponds to best quality of life.
Time Frame: At 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 7
score on a scale
  Communication | 19 (11)
  Work / Finance | 14 (24)
  Hobbies / Leisure | 25 (31)
  Physical | 28 (20)
  Psychosocial | 12 (8)

9. Secondary Outcome: Mean Quality of Life for Essential Tremor Subjects as Measured by the Quality of Life in Essential Tremor (QUEST) at 6 Months
Description: Mean quality of life will be measured by the QUEST for ET subjects at 6 months follow-up visit. The QUEST questionnaire consists of 30 items, which are rated from 0 to 4, corresponding to the frequency (from never to always). Those 30 items assess how tremor impacts a function or how it can be associated with feelings or attitudes. The 30 items contribute to five sub scales (number of items contributing to each scale in parentheses): Physical/ADL (9), Psychosocial (9), Communication (3), Hobbies/Leisure (3), and Work/Finances (6). The score on each sub scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. Maximal score of 100 indicates worse quality of life, while minimal score 0 corresponds to best quality of life.
Time Frame: At 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 7
score on a scale
  Communication | 15 (13)
  Work / Finance | 5 (14)
  Hobbies / Leisure | 20 (32)
  Physical | 41 (26)
  Psychosocial | 13 (12)

10. Secondary Outcome: Mean Duration of Programming
Description: Duration of programming at the Informity programming visit compared to the most recent programming session prior to enrollment
Time Frame: At Day 21
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single Arm
Number analyzed (Participants) | 7
minutes
  Last programming session | 76 (70)
  Informity programming session | 85 (37)

11. Secondary Outcome: Change in Therapeutic Electrical Energy Delivered (TEED) at 3 Months
Description: Change in TEED at the 3-month follow-up visit compared to baseline
Time Frame: At 3 months compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Arm/Group | Single Arm
Number analyzed (Participants) | 7
milliampere (mA)
  Baseline | 44.8 (32.7)
  3 months | 75.1 (70.1)

12. Secondary Outcome: Change in Therapeutic Electrical Energy Delivered (TEED) at 6 Months
Description: Change in TEED at the 6-month follow-up visit compared to baseline
Time Frame: At 6 months compared to baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: milliampere (mA)
Arm/Group | Single Arm
Number analyzed (Participants) | 7
milliampere (mA)
  Baseline | 44.8 (32.7)
  6 months | 76.0 (75.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=8)
Spine fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Extension malfunction (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=8)
Persistent pain, tightness, or discomfort around the implanted parts (Injury, poisoning and procedural complications) | 1 (1)
Initial jolt, or tingling stimulation (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Subjects enrolled at the experienced centers in this study already had individually tailored therapy at the baseline visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT03794661/Prot_SAP_000.pdf